CLINICAL TRIAL: NCT04731753
Title: Post Market Clinical Follow up Study to Examine Clinical Performance of the Debridement Pad Cutimed DebriClean
Brief Title: PMCF Study to Examine the Debridement Pad Cutimed DebriClean
Status: Completed | Type: Observational
Sponsor: BSN Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: BSN-C2533
Record Dates: First submitted 2021-01-18; First posted 2021-02-01 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-02

CONDITIONS: Wound
Keywords: Debridement
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group treated with study product: Subjects will undergo one mechanical debridement procedure with Cutimed DebriClean
  Interventions: Device: mechanical debridement

INTERVENTIONS:
Device: mechanical debridement — The mechanical debridement is performed using the debridement pad Cutimed DebriClean. After the pad is moistened with wound-cleansing solution, the wound is cleaned using circular movements while applying gentle pressure.

SUMMARY:
Documentation of the performance and safety of the debridement pad Cutimed DebriClean in daily clinical practice

DETAILED DESCRIPTION:
60 subjects with superficial wounds in need of debridement will undergo mechanical debridement with the study product.

Per subject, one application of the study product will be documented including photo documentation of the wound and evaluation of the wound bed condition and wound size before and after the debridement.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older with full legal competence
* Signed informed consent
* Subjects with wounds in need of debridement, especially diabetic ulcers, venous and arterial ulcers, pressure sores, postoperative wounds and wounds healing by secondary intention, superficial burns
* Superficial wound
* Minimum 30 % of the wound is covered by debris, necrosis or slough
* Wound size > 4 cm²

Exclusion Criteria:

* Subjects not willing to participate or to attend the scheduled study visit
* Known sensitivity or allergy to the product components
* Severe pain or hyperaesthesia in the wound area
* Patients who are pregnant or lactating
* Drug abuse or alcohol abuse
* Patients who participate in any other clinical study investigating drugs or medical devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with superficial wounds in need of debridement, for example diabetic ulcers, venous and arterial ulcers, pressure sores, postoperative wounds and wounds healing by secondary intention, superficial burns, the absorption of exudate, slough and dry skin flakes.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Change of wound bed condition from baseline to assessment immediately after the mechanical debridement (within one study visit) | assessed immediately before and immediately after the mechanical debridement (within one study visit)
  Percentage of wound coverage with debris/necrosis/slough Wound edge cleaned smooth Surrounding skin cleaned e.g. from skin flakes

SECONDARY OUTCOMES:
Wound size after and before wound debridement | assessed immediately before and immediately after the mechanical debridement (within one study visit)
  Wound length and wound width are measured using a wound ruler. Wound size is calculated using the formula A = length x width x π/4.
Time needed for the debridement procedure | Time is measured during the debridement procedure
  Time from start to completion of the debridement procedure in minutes
Debris/necrosis/slough absorbed by test product | assessed immediately after the mechanical debridement
  assessed by the investigator (five categories)
Structural integrity of the test product | assessed immediately after the mechanical debridement
  assessed by the investigator (e.g. change in shape, loosening of fibers, …)
Pain during the debridement procedure | assessed immediately after the debridement procedure
  Patient reported pain assessed using a visual analogue scale. If applicable, duration of pain is documented.
Adverse device effects | assessed immediately after the debridement procedure
  Discomfort, pressure, burning sensation, bleeding, and irritation of the periwound skin during or after the mechanical debridement, other adverse device effects swelling; redness

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Atkin, Dr., Principal Investigator — The University of Huddersfield
Locations (3):
- Germany (2):
  - Praxis am Stadtpark, Ahlen, North Rhine-Westphalia
  - Universitäres Herz- und Gefäßzentrum, Universitätsklinikum Hamburg-Eppendorf, Hamburg
- Pinderfields Hospital, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared. Data are needed for post market clinical follow up.